CLINICAL TRIAL: NCT06448078
Title: Comparative Evaluation of External Chest Wall Fixator Treatment Effectiveness in Patients With Rib Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gizem Kececi Ozgur, Principal investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GKOzgur
Record Dates: First submitted 2024-05-31; First posted 2024-06-07 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-08

CONDITIONS: Rib Fractures; Trauma
Keywords: rib fracture; external chest wall fixator; trauma
MeSH Terms: conditions — Rib Fractures; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Within the scope of the study, external fixator will be applied to 14 patients in the form of external bonding to the rib fracture area for 15 days, along with standard medical treatment. Standard medical treatment will be applied to 20 patients and these patients will constitute the control group.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Active Comparator): External chest wall fixator will be applied to the rib fracture area in the case group
  Interventions: Device: External chest wall fixator
- Control group (No Intervention): No intervention will be made to the control group

INTERVENTIONS:
Device: External chest wall fixator — External chest wall fixator is applied in the form of external bonding to the rib fracture area
  Arms: Case group

SUMMARY:
This study aimed to investigate the effect of external chest wall fixator on patients' pain level, complication development and hospital stay in patients with rib fractures.Patients who were admitted due to trauma and had serial rib fractures were evaluated. Standard treatment was applied to the control group. External chest wall fixator was applied to the case group in standard treatment. Pain levels of the patients, development of complications and duration of hospitalization were recorded.

DETAILED DESCRIPTION:
Basis of treatment for rib fractures is pain control and physiotherapy. External chest wall fixators may provide a new approach as part of multimodal treatment. This study aimed to investigate the effect of external chest wall fixator on patients' pain level, complication development and hospital stay in patients with rib fractures.

Patients who were admitted due to trauma and had serial rib fractures were evaluated. There were 14 patients in case group and 20 in control group. Standard treatment was applied to the control group. External chest wall fixator was applied to the case group in addition to standard treatment. Pain levels of the patients, development of complications and duration of hospitalization were recorded. Pain levels of the patients were evaluated using the Visual Analogue Scale and the pain level was scored between 0 and 10.

ELIGIBILITY:
Inclusion Criteria:

* Patients with serial rib fractures after trauma
* Patients without extrathoracic pathology

Exclusion Criteria:

* Patients with less than 3 rib fractures
* Patients with extrathoracic injuries
* Patients with bilateral rib fractures
* Patients with flail chest
* Patients with hemothorax or pneumothorax requiring drainage with tube thoracostomy at first admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Kececi Ozgur, MD, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Medicine, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data of the study will be shared if requested from the authors
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: The responsible researcher can be contacted via e-mail

REFERENCES:
- [Background] Lee Y, Lee SH, Kim C, Choi HJ. Comparison of the effectiveness in pain reduction and pulmonary function between a rib splint constructed in the ER and a manufactured rib splint. Medicine (Baltimore). 2018 May;97(21):e10779. doi: 10.1097/MD.0000000000010779. PMID 29794759
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614
- [Background] Martin TJ, Eltorai AS, Dunn R, Varone A, Joyce MF, Kheirbek T, Adams C Jr, Daniels AH, Eltorai AEM. Clinical management of rib fractures and methods for prevention of pulmonary complications: A review. Injury. 2019 Jun;50(6):1159-1165. doi: 10.1016/j.injury.2019.04.020. Epub 2019 Apr 22. PMID 31047683
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Case Group | Control Group
Started | 14 | 20
Completed | 14 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Case Group | Control Group | Total
Number analyzed (Participants) | 14 | 20 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.50 (19.55) | 52.50 (13.80) | 55.38 (16.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 10 | 16 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 14 | 20 | 34

OUTCOME MEASURES:

1. Primary Outcome: Pain Level
Description: Pain level of patients on the 10th day, 1st month and 3rd month (Visual Analogue Pain Scale (VAS) will be used to assess pain level.Pain level will be scored between 1 and 10.Higher scores represent worse outcomes.)
Time Frame: 3 months
Population: first month pail level
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 14 | 20
score on a scale | 1.79 (0.80) | 2.85 (1.53)

2. Primary Outcome: Complications
Description: Number of participants who developed complications
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 14 | 20
Participants | 2 | 8

3. Primary Outcome: Hospital Stay
Description: Duration of hospital stay of patients (days)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 14 | 20
day | 2.00 (0.784) | 2.70 (0.979)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Case Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/20
Other Adverse Events (participants affected / at risk) | 0/14 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT06448078/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT06448078/ICF_001.pdf